CLINICAL TRIAL: NCT04561661
Title: A Randomized Comparison Between Percutaneous Pinning and Non-surgical Management of Proximal Phalangeal Fractures
Brief Title: Percutaneous Pinning vs Orthosis and Early Mobilization
Acronym: POEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Wilcke, MD, Phd, Associate prof, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Frakturstudien
Record Dates: First submitted 2020-09-14; First posted 2020-09-23 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Hand Injuries; Finger Fracture
MeSH Terms: conditions — Hand Injuries | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conservative treatment (Active Comparator): Fracture treated with closed reduction, custom made orthosis and early mobilization.
  Interventions: Procedure: Conservative treatment
- Surgery (Active Comparator): Fractures treated with closed reduction, percutaneous pinning (k-wires) and plaster.
  Interventions: Procedure: Percutaneous pinning

INTERVENTIONS:
Procedure: Percutaneous pinning — Closed reduction, percutaneous pinning and plaster
  Arms: Surgery
Procedure: Conservative treatment — Closed reduction, custom made orthosis and early mobilization
  Arms: Conservative treatment

SUMMARY:
This study aims at investigating if splinting and early mobilization is a better method, regarding range of motion, for treating fractures of the base phalanx of the fingers compared to surgery with pinning. This will be achieved through a randomised clinical trial comparing the two methods.

DETAILED DESCRIPTION:
Proximal phalangeal fractures of the hand are very common and affect patients of all ages. . Most fractures heal without complications but these injuries can result in impaired hand function and prolonged inability to work and perform activities of daily living. If there is a dislocation that cannot easily be repositioned to a stable position, surgery might be required. Surgery is often performed with percutaneous pinning and immobilisation in plaster for 4 weeks. Good results of non-surgical treatment with a splint that allows immediate mobilization of the interphalangeal joints has been reported. This study will compare these two methods for treating fractures of the base phalanx of the fingers. Recruited patients will be randomized to one of the two treatment arms: 1. surgery with pinning 2. conservative treatment with a splint. Primary outcome is total active range of motion in the affected finger at 3, 6 months and 1 , 3 years. Secondary outcomes are number of sick days and various patient related outcome measures.

ELIGIBILITY:
Inclusion Criteria:

-Fractures of the base phalanx of digit 2-5 in the hand.

Exclusion Criteria:

* Fracture older than 2 weeks.
* More than 25° of sagittal plane and/or 10° lateral angulation after reposition.
* Intra-articular step >1mm.
* Associated fractures in other bones (i e metacarpals, middle and distal phalanges) and/or tendon and nerve injuries in any finger.
* Open fractures.
* Patient age <18 years.
* Inability to co-operate with the follow-up protocol (i.e. language difficulties, severe psychiatric disorder, cognitive impairment, drug addiction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
TAM (Total active range of motion) | 3 months
  Total active range of motion measured in degrees of the affected finger.
TAM (Total active range of motion) | 6 months
  Total active range of motion measured in degrees of the affected finger.
TAM (Total active range of motion) | 1 year
  Total active range of motion measured in degrees of the affected finger.
TAM (Total active range of motion) | 3 years
  Total active range of motion measured in degrees of the affected finger.

SECONDARY OUTCOMES:
Number of sick days | 3 months
  Number of sick days from the intervention until full return to work.
Patient related outcome measure DASH | 3, 6 months and 1 and 3 years
  Disability of the Arm, Shoulder and Hand score (DASH). 0 points means no disability and 100 maximum disability.
Patient related outcome measure HADS | 3, 6 months and 1 and 3 years
  Hospital Anxiety and Depression Scale (HADS). The score is consists of one depression scale from 0 to 21, where 0 is no signs of depression and one anxiety scale from 0 to 21, where 0 means no anxiety.
Patient related outcome measure EQ-5D | 3, 6 months and 1 and 3 years
  EuroQols quality of life index. Consists of an index based on the questionnaire where 0 means death and 1 means full quality of life and one visual analog scale 0-100 where patients rate their health from bad (0) to excellent (100).
Patient related outcome measure HQ-8 | 3, 6 months and 1 and 3 years
  HQ-8 is a questionnaire specifically for hand injuries. Each question gives a score 0-100, where 0 means no problems and 100 means worst imaginable problem.
Grips strength | 3, 6 months and 1 and 3 years
  Measured in kilograms (JAMAR)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna von Kieseritzky, MD PhD, Study Director — Karolinska Institutet
Locations (1):
- Dept Hand Surgery, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No